CLINICAL TRIAL: NCT03116906
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 685509 in Healthy Male Subjects
Brief Title: Safety and Tolerability of BI 685509 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1366.3; 2014-004540-35 (EudraCT Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-17 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 685509 (Experimental): multiple rising doses of BI 685509
  Interventions: Drug: BI 685509
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 685509 — to be given for a total of up to 15 days
  Arms: BI 685509
Drug: Placebo — to be given for a total of up to 15 days
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 685509 in healthy male subjects following oral administration of multiple rising doses.

Secondary objectives are the exploration of the pharmacokinetics (PK), dose proportionality, the attainment of steady state, as well as investigation of linearity and pharmacodynamics (PD) of BI 685509 after multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP (Blood Pressure), PR (Pulse Rate)), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* Body Mass Index of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP (Blood Pressure), PR (Pulse Rate), or ECG (Electrocardiogram)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 60 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm (beats per minute)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during in-house confinement
* Alcohol abuse (consumption of more than 24 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related Adverse Events | 5 weeks

SECONDARY OUTCOMES:
AUC tau,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval tau after administration of the first dose) [AUC tau,1 will be AUC0-24 for QD] | up to 24 hours
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours
AUC tau,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval tau) [AUC tau,ss will be AUC0-12,ss for bid and AUC0-24,ss for QD] | up to 408 hours
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval tau) | up to 408 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong D, Seitz F, Bauer V, Giessmann T, Schulze F. Safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 685509, a soluble guanylyl cyclase activator, in healthy volunteers: Results from two randomized controlled trials. Naunyn Schmiedebergs Arch Pharmacol. 2024 Oct;397(10):8101-8116. doi: 10.1007/s00210-024-03165-w. Epub 2024 May 24. PMID 38789635